CLINICAL TRIAL: NCT03478501
Title: Assisting in Informing Decisions in Emergency Departments: (ED-AID) Study
Brief Title: Assisting in Decisions in Emergency Departments: (ED-AID) Study
Acronym: ED-AID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Denver Health and Hospital Authority (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-2299; R34MH113539-01 (NIH)
Record Dates: First submitted 2018-03-01; First posted 2018-03-27 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Suicide; Emergencies
Keywords: firearm; lethal means; decision aid
MeSH Terms: conditions — Suicide; Emergencies | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision Aid Group (Experimental): Participants randomized to this arm will view the decision aid on a tablet in the emergency department.
  Interventions: Behavioral: Decision Aid
- Control Group (No Intervention): Participants randomized to this arm will be asked to review general suicide prevention information on a tablet in the emergency department.

INTERVENTIONS:
Behavioral: Decision Aid — This intervention is a tablet based Lethal Means Decision Aid with proposed use to augment lethal means counseling in emergency departments for patients at risk of suicide.
  Arms: Decision Aid Group

SUMMARY:
This study will test a patient decision aid about safe firearm storage during suicidal crisis. The investigators hypothesize that participants with higher quality decisions after the decision aid will be more likely to change their firearm storage to reduce access during the time of crisis.

DETAILED DESCRIPTION:
Limiting access to a firearms during suicidal crisis can save lives. This study will test a patient decision aid about safe firearm storage during crisis. The investigators will enroll 60 adult emergency department patients being evaluated for suicidal risk and have at least one firearm at home. If available, the investigators will also enroll a family member or friend. Participants will randomly receive one of two things: the decision aid or general suicide prevention information. A week later, the investigators will call participants to see how both groups choose to store their firearms. This trial tests the acceptability of the decision aid, effects on decision making, effect on home storage, effect on suicide outcomes, and feasibility of a larger trial. The investigators hypothesize that participants with higher quality decisions after the decision aid will be more likely to change their firearm storage to reduce access during the time of crisis; should the pilot demonstrate feasibility, in a subsequent larger trial this hypothesis would be tested directly.

ELIGIBILITY:
Inclusion Criteria:

* Being evaluated in the emergency department for suicidal ideation/suicide attempt
* Deemed medically stable by ED physician
* Age greater than or equal to 18 years old
* Able and willing to have telephone follow up at 1 week
* Report at least one firearm in the home

Exclusion Criteria:

* Unable to participate medically or cognitively (e.g. sustained altered level of consciousness, hostility, psychosis, sexual assault victim, severe vomiting or pain)
* Currently in legal custody
* Live in group home or other supervised custody
* Already enrolled

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Acceptability of Lethal Means Decision Aid | Baseline
  This will be assessed using the Ottawa Acceptability Questionnaire that captures the patient's feedback on the design, presentation, quality, and information presented in the decision aid through both survey and open ended questions. Questions include likert scale responses (range of responses are specific to each question's content). There are also a series of yes/no/don't know questions related to content presented. Each "no" response asks the participant to elaborate in an open ended response. The participant also has the ability to provide general feedback in open ended feedback format. There are no subscales to this measure.
Decision Making Quality in Emergency Department (ED) | Baseline
  The Decisional Conflict Scale (DCS), low literacy 10 item scale, measures decision quality, uncertainty, personal perceptions and satisfaction. A total score is computed through sum of items 1-10 (Yes=1; unsure=2; no=4) divided by 10, and multiplied by 25. Scores range from 0 (no decision conflict) to 100 (extreme decision conflict). The sum of items 1, 2, 3, divided by 3 and multiplied by 25 is the informed decision subscale (1 extremely informed) to 100 extremely uninformed). The sum of items 4 and 5, divided by 2 and multiplied by 25 is the values clarity (0 feels extremely clear to 100 feels extremely unclear). The sum of items 9 and 10, divided by 2 and multiplied by 25 is the uncertainty subscale (0 feels extremely certain about best choice to 100 feels extremely uncertain about best choice). The sum of items 6, 7, 8, divided by 3 and multiplied by 25 is the support subscale (0 feels extremely supported in decision making to 100 feels extremely unsupported in decision making).
Home Firearm Storage | Baseline and 1 week follow up
  At both baseline and one week follow up, participants will complete a study specific survey that asks about how they currently store their firearms or current plans to change how they store their firearms to measure change in storage.
Decision Making Quality - Follow up | 1 week follow up
  The Decisional Conflict Scale (DCS), low literacy 10 item scale, measures decision quality, uncertainty, personal perceptions and satisfaction. A total score is computed through sum of items 1-10 (Yes=1; unsure=2; no=4) divided by 10, and multiplied by 25. Scores range from 0 (no decision conflict) to 100 (extreme decision conflict). The sum of items 1, 2, 3, divided by 3 and multiplied by 25 is the informed decision subscale (1 extremely informed) to 100 extremely uninformed). The sum of items 4 and 5, divided by 2 and multiplied by 25 is the values clarity (0 feels extremely clear to 100 feels extremely unclear). The sum of items 9 and 10, divided by 2 and multiplied by 25 is the uncertainty subscale (0 feels extremely certain about best choice to 100 feels extremely uncertain about best choice). The sum of items 6, 7, 8, divided by 3 and multiplied by 25 is the support subscale (0 feels extremely supported in decision making to 100 feels extremely unsupported in decision making).
Suicidal Ideation and Behavior at One Month | 1 month post baseline
  While this pilot trial is not powered to detect a change in mental health outcomes, as part of the feasibility for a larger trial, the investigators will attempt to track suicide attempts and outcomes through medical record chart review.
Suicidal Ideation and Behavior at Three Months | 3 months post baseline
  While this pilot trial is not powered to detect a change in mental health outcomes, as part of the feasibility for a larger trial, the investigators will attempt to track suicide attempts and outcomes through medical record chart review.
Vital Statistics (Suicide death) | 3 months post baseline
  While this pilot trial is not powered to detect a change in suicide outcomes, as part of the feasibility for a larger trial, the investigators will attempt to track suicide death outcomes through state vital statistics reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Betz, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Hospital, Aurora, Colorado
  - Memorial Hospital, Colorado Springs, Colorado
  - Denver Health, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Betz ME, Knoepke CE, Simpson S, Siry BJ, Clement A, Saunders T, Johnson R, Azrael D, Boudreaux ED, Omeragic F, Adams LM, Almond S, Juarez-Colunga E, Matlock DD. An Interactive Web-Based Lethal Means Safety Decision Aid for Suicidal Adults (Lock to Live): Pilot Randomized Controlled Trial. J Med Internet Res. 2020 Jan 29;22(1):e16253. doi: 10.2196/16253. PMID 32012056

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT03478501/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT03478501/ICF_001.pdf